CLINICAL TRIAL: NCT01790542
Title: Assessment of Complementary Feeding of Canadian Infants
Acronym: Infant Feeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: H2011:166
Record Dates: First submitted 2013-02-06; First posted 2013-02-13 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2014-07

CONDITIONS: Generation of Reactive Oxygen Species; Intestinal Inflammation
Keywords: Iron; Intestinal inflammation; ROS
MeSH Terms: interventions — Fruit; Meat

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Other): Iron fortified cereal
  Interventions: Other: Iron fortified cereal
- B (Other): Iron fortified cereal with fruit
  Interventions: Other: Iron fortified cereal with fruit
- C (Other): Meat
  Interventions: Other: Meat

INTERVENTIONS:
Other: Iron fortified cereal — Infants will be assigned to one of the three interventions: A (iron fortified cereal), B (iron fortified cereal with fruit), C (Meat)
  Other Names: Infant feeding
  Arms: A
Other: Iron fortified cereal with fruit
  Arms: B
Other: Meat
  Arms: C

SUMMARY:
With the recent recommendation from Health Canada to extend exclusive breast-feeding to 6 months of age there has arisen concern about what is the best solid food to introduce at that time. Traditionally solids were introduced in Canada at 4-6 months and usually iron-fortified rice cereal was the first food of choice. New recommendations from Health Canada include meat as a potential first food as well as other iron fortified foods. This has lead to uncertainty of both public health officials and parents about the optimal introduction and choice of solids after exclusive breastfeeding.

In addition to meeting iron needs with the first solid food choice, the investigators are concerned about the possible generation of reactive oxygen species (ROS) in the gut of the infant fed traditional iron fortified cereals. Infant cereals are fortified at 25-30 mg iron per 100 g dry-weight. Absorption of the non-heme electrolytic iron ranges from 5-10% so that most of the residual iron enters the colon. Normally excess iron is sequestered by a variety of mechanisms in the body, but there is no such system for the sequestering of iron in the gut lumen. The investigators have shown that providing iron supplements to adults where the majority of the iron is unabsorbed passes through the digestive tract can lead to the generation of ROS in the colon. These effects are seen in adults receiving 1 mg/kg/day supplemental iron. By 5-6 months of age infants consuming iron fortified cereals will receive the same dose and are likely producing ROS in their digestive tract. This may cause inflammation and make infants more susceptible to disease. The investigators think that meats and infant cereals with phenolic antioxidants available from fruits will likely reduce the generation of ROS in vivo. Therefore the investigators wish to determine if traditional and newly recommended first foods are safe from a free radical and inflammatory perspective.

HYPOTHESES:

1. Consumption of infant cereals with iron will increase ROS generation in the gut
2. Consumption of infant cereals with iron and fruit will decrease ROS in the gut
3. Consumption of meat will not generate ROS
4. Consumption of iron fortified cereals or meat will maintain iron status during infancy

ELIGIBILITY:
Inclusion Criteria:

* Full term infant
* Birth weight more than 2500g
* Absence of any medical conditions

Exclusion Criteria:

* Consumption of more than 200ml formula

Max Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 87 (Actual)
Dates: Start 2012-12; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in production of ROS | Before introduction of study food and 2-3 weeks after introduction of study food
  Production of reactive oxygen species

SECONDARY OUTCOMES:
Change in Microbiome | Before introduction of study food and 2-3 weeks after introduction of study food
  Microflora of term infants before and after the introduction of solids
Change in Fecal Calprotectin | Before introduction of study food and 2-3 weeks after introduction of study food
  Inflammatory marker
Fecal non heme iron production | Before introduction of study food and 2-3 weeks after introduction of study food
  Non heme iron founded in infant cereal is less absorbed, remains in the gut, and excreted in the feces.
Dietary iron intake from first complementary food | 3 days dietary record
Micro and Macro nutrient intake of breastfed infants from first complementary food | 3 days dietary record

OTHER OUTCOMES:
Change in 8OH-deoxyguanosine | Before introduction of study food and 2-3 weeks after introduction of study food
  Oxidative stress marker in the urine
Change in F2 Isoprostane | Before introduction of study food and 2-3 weeks after introduction of study food
  Oxidative stress marker in the urine

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

REFERENCES:
- [Derived] Qasem W, Azad MB, Hossain Z, Azad E, Jorgensen S, Castillo San Juan S, Cai C, Khafipour E, Beta T, Roberts LJ 2nd, Friel J. Assessment of complementary feeding of Canadian infants: effects on microbiome & oxidative stress, a randomized controlled trial. BMC Pediatr. 2017 Feb 14;17(1):54. doi: 10.1186/s12887-017-0805-0. PMID 28196533
- See also: Study Information — http://www.facebook.com/pages/Assessment-of-Complementary-Feeding-of-Canadian-Infants-Study/529407130412012